CLINICAL TRIAL: NCT06111131
Title: A Randomized Controlled Trial to Demonstrate the Ancora-SB Overtube Complete Positioning and Optical Visualization During Endoscopic Procedures for Diagnosis and Treatment in the Small Intestine
Brief Title: Ancora-SB Overtube Complete Positioning and Optical Visualization During Endoscopic Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aspero Medical, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASPE-CLIN-2022-01
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Small Bowel Disease
Keywords: Small Intestine

STUDY DESIGN:
Intervention Model Description: This is a double-blind randomized 1:1 controlled post-market study; the investigator and the subject will be blind to the device. A qualified staff member will assist the endoscopist by performing the preparation, insertion, and removal of the device the subject was randomized to, to ensure the investigator is blinded. The shaft and handle end of the Ancora-SB overtube will be the same as the Olympus ST-SB1 overtube.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ancora-SB Overtube (Active Comparator): Enteroscopy with Ancora-SB Balloon Overtube
  Interventions: Device: Enteroscopy
- Olympus ST-SB1 Overtube (Active Comparator): Enteroscopy with Olympus ST-SB1 Overtube
  Interventions: Device: Enteroscopy

INTERVENTIONS:
Device: Enteroscopy — A procedure that uses a specially equipped endoscope to examine the small intestine lining. An enteroscopy uses an endoscope, a tube with a light and camera on the end and the endoscope, in the case of this study, is equipped with a single balloon overtube to advance the scope deeper into the small intestine, to reach the middle third of the small bowel.

SUMMARY:
Demonstrate superiority of the Aspero Medical Ancora-SB balloon Overtube compared to the Olympus ST-SB1 Balloon Overtube.

DETAILED DESCRIPTION:
The study objective, demonstrate superiority of the Aspero Ancora-SB balloon overtube compared to the Olympus ST-SB1 Balloon Overtube, is necessary for adoption by clinicians. Broad adoption is expected to improve procedure success rates, reduce time to diagnosis or treatment (thereby, improving patient outcomes), and reduce the burden and costs of care for patients, providers, and insurers. Investigators propose to recruit patients scheduled for enteroscopy and use capsule endoscopy to identify patients with lesions in the middle third of the small bowel. The primary outcome of interest is success in identifying the lesion, which indicates sufficient balloon control to reach and visualize the site.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent;
2. Subject meets the minimal safety criteria for single balloon enteroscopy: ASA Class I, II, or III;11
3. ≥ 18 years of age to ≤ 90 years of age;
4. Video capsule endoscopy identified lesions in the middle third of the small bowel;
5. Willing and able to comply with all study procedures and follow-up.

Exclusion Criteria:

1. History of gastric bypass or related procedures;
2. History of foregut and/or midgut surgery;
3. Pathology identified by video capsule is in the proximal 1/3 of the bowel;
4. Pathology identified by video capsule is in the distal 1/3 of the bowel;
5. Anticoagulant and antiplatelet therapy that cannot be stopped for the enteroscopy;
6. Capsule endoscopy did not show clear visualization of pathology in the middle small bowel;
7. Inability to tolerate the investigator's method of sedation that is the standard of care;
8. Any previous small bowel surgery, or anastomosis, that caused extensive adhesions and/or altered anatomy;
9. Allergy to any medications or product used in the endoscopic procedure where the severe allergic reaction cannot be prevented with pre-medication;
10. Pregnancy;
11. Life expectancy < six (6) months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Device Superiority | Enteroscopy Procedure
  Demonstrate superiority of the Aspero Medical Ancora-SB balloon Overtube compared to the Olympus ST-SB1 Balloon Overtube. Superiority of the Ancora-SB Balloon Overtube will be demonstrated if it achieves a success rate of ≥75% compared to a success rate of 50% with the Olympus ST-SB1 Balloon Overtube.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Cedars Sinai, Los Angeles, California
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No